CLINICAL TRIAL: NCT02616627
Title: Association Between DXA Results and the Complications, Clinical Courses and Outcomes in Chronic Dialysis Patients
Status: Recruiting | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201505154RINB
Record Dates: First submitted 2015-11-25; First posted 2015-11-30 (Estimated); Last update posted 2022-05-04 (Actual); Status verified 2022-05

CONDITIONS: Chronic Kidney Disease Requiring Chronic Dialysis; Osteoporosis
Keywords: bone mineral density; chronic dialysis; end-stage renal disease; body composition analysis; sarcopenia
MeSH Terms: conditions — Osteoporosis; Kidney Failure, Chronic; Sarcopenia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- chronic dialysis: Patient enrolled at the National Taiwan University Hospital Jinshan branch

SUMMARY:
Aims:

1. To determine whether BMD and muscle mass were associated with fractures and other adverse events in dialysis patients.
2. To explore the effects of the interactions among FGF23, calcium, phosphate, PTH and vitamin D on low bone mineral density and sacropenia in dialysis patients.

Method:

In this study, the investigators plan to use DXA to screen for BMD, relevant novel bone microstructure parameters, and body composition in chronic dialysis patients. Also, the investigators plan to use blood testing to measure the blood level of FGF23, calcium, phosphate, PTH and vitamin D. The investigators conduct a prospectively follow up program for these participants to evaluate clinical courses and outcomes. Patients will receive DXA (including BMD and body composition) tests and blood work at baseline and one-year. Muscle power and physical performance will be measured at baseline, 6 months and one-year.

DETAILED DESCRIPTION:
Background:

Several large-scale studies enrolling CKD patients discovered that low BMD is still an important risk factor for developing fragility fractures, while chronic dialysis patients are reported to have 4 to5 fold higher risk of fracture compared to general population. However, the relationship between bone mineral density (BMD) by dual-energy X-ray absorptiometry (DXA) and fracture and other adverse events in patients with CKD patients is still unclear. In addition, declining of renal function could affect the normal physiological regulating of blood levels of calcium, phosphate, fibroblast growth factor 23 (FGF23), parathyroid hormone (PTH), and vitamin D, which could influence the bone mineral density of chronic dialysis patients. Recently, it is well known that serum FGF23 is already elevated at the early stage of CKD patients and independently related to CKD. However, there are a limited number of reports indicate that the effects of the interactions among FGF23, calcium, phosphate, PTH and vitamin D on low bone mineral density and sacropenia in CKD patients.

Aims:

1. To determine whether BMD by DXA was associated with fractures and other adverse events in dialysis patients.
2. To explore the effects of the interactions among FGF23, calcium, phosphate, PTH and vitamin D on low bone mineral density and sacropenia in dialysis patients.

Method:

In this study, the investigators plan to use DXA to screen for BMD, relevant novel bone microstructure parameters, and body composition in chronic dialysis patients. Also, the investigators plan to use blood testing to measure the blood level of FGF23, calcium, phosphate, PTH and vitamin D. The investigators conduct a prospectively follow up program for these participants to evaluate clinical courses and outcomes.

Patient characteristics

Inclusion Criteria:

1. Age >20 years and one of the below
2. Chronic hemodialysis
3. Chronic peritoneal dialysis

Exclusion Criteria:

get pregnant or planning a pregnancy

Anticipated results:

1. The investigators expect that results and findings discovered from this study could show the effects of interactions of FGF23, calcium, phosphate, PTH and vitamin D on low bone mineral density and sacropenia in CKD patients, which should be an important step on improving clinical decision for osteoporosis and fracture risk in renal dialysis patients.
2. Publishing results in an academic journal.

ELIGIBILITY:
Patient characteristics

Inclusion Criteria:

1. Age >20 years and one of the below
2. Chronic hemodialysis
3. Chronic peritoneal dialysis

Exclusion Criteria:

1. get pregnant or planning a pregnancy

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chronic Kidney Disease Requiring Chronic Dialysis
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2015-09; Primary Completion 2021-03 (Actual); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Bone mineral density by DXA, | one year
  Change of BMD between baseline and one year was measured

SECONDARY OUTCOMES:
Blood tests | one year
  Change of baseline and one year value of various blood tests mentioned in the summary
Sarcopenia | baseline, 6 month and one year
  Changes of saropenia percentage at 6 month and one year compared to baseline assessments. 3 measures were used, muscle mass, grip strength, and walking speed

CONTACTS AND LOCATIONS:
Overall Officials: Ding-Cheng Chan, MD, PhD, Principal Investigator — National Taiwan University Hospital, Chutung branch
Locations (1):
- National Taiwan University Hospital, Chutung branch, Hsinchu, Taiwan